CLINICAL TRIAL: NCT04184154
Title: Vaginal Dilatators and Moisturizers Use and Sexual Quality of Life of Patients With Gynecologic Cancer Treated With Brachytherapy.
Brief Title: Sexual Quality of Life of Patients With Gynecologic Cancer Treated With Brachytherapy.
Acronym: Gyn&Co
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: ICM-URC 2017/14
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2019-12

CONDITIONS: Pelvic Cancer; Cervical Cancer
Keywords: cervical and endometrial cancer; brachytherapy; patient education program; sexual quality of life; vaginal stenosis; patient-reported outcomes
MeSH Terms: conditions — Pelvic Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — The self-questionnaire of 104 questions collected personal and socio-demographics data, global and sexual quality of life characteristics (European Organisation for Research and Treatment of Cancer [EORTC] quality of life questionnaires: QLQ-C30 and gynecologic and cervical cancer specific-questionnaire QLQ-CX24), vaginal dilatators and moisturizers use, and barriers and facilitators of their use. Clinical data were extracted from the patients' medical files. Vaginal stenosis was evaluated at 6 weeks after the end of brachytherapy and after 1-year follow-up by in-town gynecologists or in our Institute, and censored in case of complete vaginal obliteration

SUMMARY:
Gynecologic cancer treatments (chemoradiotherapy, brachytherapy and surgery) greatly impact patients' sexual quality of life (QoL). Use of the vaginal dilators may reduce vaginal stenosis. Since 2011, our "Gyn and Co LR" patient education program aims to optimize early care of sexual disorders following treatment of cervical and endometrial cancer.

DETAILED DESCRIPTION:
Pelvic cancer accounts for 38,000 cancer cases in France; among them, 15,500 are gynecologic, i.e. endometrial, ovarian, cervical, vaginal and vulval. In 2017, 8,367 new endometrial cancer cases were reported in France1. Endometrial cancer mostly affects women who already underwent menopause; indeed, the median age at diagnosis is 68 years. Cervical cancer is less frequent, with 2,835 new cases reported in France in 2017, but affects younger women. The incidence peak is reported at 40 years, with a median age at death of around 50 years.

The standard of care for cervical cancer combines chemoradiotherapy with utero-vaginal brachytherapy, followed or not with surgery. For endometrial cancer, post-operative vaginal brachytherapy is recommended for intermediate-risk tumors or following radiotherapy for high-risk patients. However, in both cancer localizations, the combination of external radiation and brachytherapy induces numerous adverse effects affecting the patients' overall and sexual quality of life. Digestive, urinary and sexual disorders reported include abdominal pain, incontinence, cystitis, dyspareunia, vaginal irritation, pain during intercourse. A major adverse effect reported is reduction of vaginal elasticity together with vaginal shrinking (shorter and tighter vagina), up to vaginal stenosis. The EMBRACE study showed in 630 patients with locally-advanced cervical cancer a grade ≥ 2 vaginal stenosis rate of 21% at 2 years. A study reported that among sexually active women, 54% were not satisfied or little satisfied with their sexual activity; about 50% women also reported vaginal dryness and more than 40% pain during penetration. The EMBRACE study reported in locally-advanced cervical cancer patients the persistence of treatment-related symptoms, diarrhea, menopausal symptoms, peripheral neuropathy and sexual functioning problems two years after diagnosis. Vaginal dryness, hot flashes and pain at penetration were reported up to 5 to 10 years after diagnosis in cancer survivors as compared with controls in a case-control study. In endometrial cancer patients, a long-term analysis of the PORTEC-2 study reported vaginal dryness, short or narrow vagina and pain during intercourse at 7 years after treatment.

Studies in psycho-oncology or nursing care have assessed the impact of these disorders and are bringing up some solutions, among which use of vaginal dilators to prevent vaginal stenosis and improve sexual quality of life. International guidelines were issued on the use of vaginal dilators by these patients. Both guidelines and studies assessing patient education interventions to increase the patients' use of the vaginal dilators concluded on the possible benefit of educational programs stenosis prevention. Some programs well integrated in the patients' care pathway have been published. Early interventions starting as soon as the disease announcement consult with the radiation oncologist are still needed to improve vaginal stenosis prevention and the patients' sexual quality of life.

In this context, the investigator have initiated, for the first time in France, the "Gyn and Co LR" patient education program, approved by the Regional Health Agency. This program, fully integrated in the patients' care pathway, aimed to optimize an early care of sexual disorders and prevent vaginal stenosis in patients treated with brachytherapy for cervical or endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cervical or endometrial cancer, stage I to III who received brachytherapy at the ICM between January 2014 and December 2015.
* Age ≥ 18 years
* Patient who agreed to follow an therapeutic education program during the brachytherapy treatment
* Patient who agreed, after receiving information, to participate to the study

Exclusion Criteria:

* Patient who refused to follow the therapeutic education care program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the study is composed of all patients who followed the ETP curietherapy program between January 2014 and December 2015; this potentially represents372 patients.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Socio-demographics characteristics of patients who followed the "Gyn and Co LR" education program | 1 day
  Quality of life questionnaire: EORTC-QLQ-C30, EORTC QLQ-CX24
Clinical characteristics of patients who followed the "Gyn and Co LR" | 1 day
  Quality of life questionnaire: EORTC-QLQ-C30, EORTC QLQ-CX24

SECONDARY OUTCOMES:
Rate of vaginal dilatators and moisturizers use | 1 day
  Auto questionnaire
Vaginal stenosis prevalence | 1 day
  Clinical data from the patient medical file
Urinary or sexual adverse effects | 1 day
  Clinical data from the patient medical file
Patients' overall and sexual quality of life | 1 day
  Sexual quality of life questionnaire:EORTC QLQ-CX24

CONTACTS AND LOCATIONS:
Overall Officials: Christine KERR, MD, Study Chair — Institut Régional du Cancer de Montpellier
Locations (1):
- Institut Régional du Cancer de Montpellier, Montpellier, Occ, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Potter R, Tanderup K, Kirisits C, de Leeuw A, Kirchheiner K, Nout R, Tan LT, Haie-Meder C, Mahantshetty U, Segedin B, Hoskin P, Bruheim K, Rai B, Huang F, Van Limbergen E, Schmid M, Nesvacil N, Sturdza A, Fokdal L, Jensen NBK, Georg D, Assenholt M, Seppenwoolde Y, Nomden C, Fortin I, Chopra S, van der Heide U, Rumpold T, Lindegaard JC, Jurgenliemk-Schulz I; EMBRACE Collaborative Group. The EMBRACE II study: The outcome and prospect of two decades of evolution within the GEC-ESTRO GYN working group and the EMBRACE studies. Clin Transl Radiat Oncol. 2018 Jan 11;9:48-60. doi: 10.1016/j.ctro.2018.01.001. eCollection 2018 Feb. PMID 29594251
- [Background] Colombo N, Creutzberg C, Amant F, Bosse T, Gonzalez-Martin A, Ledermann J, Marth C, Nout R, Querleu D, Mirza MR, Sessa C; ESMO-ESGO-ESTRO Endometrial Consensus Conference Working Group. ESMO-ESGO-ESTRO Consensus Conference on Endometrial Cancer: Diagnosis, Treatment and Follow-up. Int J Gynecol Cancer. 2016 Jan;26(1):2-30. doi: 10.1097/IGC.0000000000000609. PMID 26645990
- [Background] Shisler R, Sinnott JA, Wang V, Hebert C, Salani R, Felix AS. Life after endometrial cancer: A systematic review of patient-reported outcomes. Gynecol Oncol. 2018 Feb;148(2):403-413. doi: 10.1016/j.ygyno.2017.11.007. Epub 2017 Nov 14. PMID 29150143
- [Background] Pfaendler KS, Wenzel L, Mechanic MB, Penner KR. Cervical cancer survivorship: long-term quality of life and social support. Clin Ther. 2015 Jan 1;37(1):39-48. doi: 10.1016/j.clinthera.2014.11.013. PMID 25592090
- [Background] Zomkowski K, Toryi AM, Sacomori C, Dias M, Sperandio FF. Sexual function and quality of life in gynecological cancer pre- and post-short-term brachytherapy: a prospective study. Arch Gynecol Obstet. 2016 Oct;294(4):833-40. doi: 10.1007/s00404-016-4099-5. Epub 2016 Apr 27. PMID 27117556
- [Background] Greimel ER, Winter R, Kapp KS, Haas J. Quality of life and sexual functioning after cervical cancer treatment: a long-term follow-up study. Psychooncology. 2009 May;18(5):476-82. doi: 10.1002/pon.1426. PMID 18702067
- [Background] Huffman LB, Hartenbach EM, Carter J, Rash JK, Kushner DM. Maintaining sexual health throughout gynecologic cancer survivorship: A comprehensive review and clinical guide. Gynecol Oncol. 2016 Feb;140(2):359-68. doi: 10.1016/j.ygyno.2015.11.010. Epub 2015 Nov 7. PMID 26556768
- [Background] Wilmoth MC. Sexuality: a critical component of quality of life in chronic disease. Nurs Clin North Am. 2007 Dec;42(4):507-14; v. doi: 10.1016/j.cnur.2007.08.008. PMID 17996752
- [Background] Bergmark K, Avall-Lundqvist E, Dickman PW, Henningsohn L, Steineck G. Vaginal changes and sexuality in women with a history of cervical cancer. N Engl J Med. 1999 May 6;340(18):1383-9. doi: 10.1056/NEJM199905063401802. PMID 10228188
- [Background] Bruner DW, Lanciano R, Keegan M, Corn B, Martin E, Hanks GE. Vaginal stenosis and sexual function following intracavitary radiation for the treatment of cervical and endometrial carcinoma. Int J Radiat Oncol Biol Phys. 1993 Nov 15;27(4):825-30. doi: 10.1016/0360-3016(93)90455-5. PMID 8244811
- [Background] Brand AH, Bull CA, Cakir B. Vaginal stenosis in patients treated with radiotherapy for carcinoma of the cervix. Int J Gynecol Cancer. 2006 Jan-Feb;16(1):288-93. doi: 10.1111/j.1525-1438.2006.00348.x. PMID 16445647
- [Background] Hofsjo A, Bergmark K, Blomgren B, Jahren H, Bohm-Starke N. Radiotherapy for cervical cancer - impact on the vaginal epithelium and sexual function. Acta Oncol. 2018 Mar;57(3):338-345. doi: 10.1080/0284186X.2017.1400684. Epub 2017 Nov 15. PMID 29140150
- [Background] Kirchheiner K, Nout RA, Lindegaard JC, Haie-Meder C, Mahantshetty U, Segedin B, Jurgenliemk-Schulz IM, Hoskin PJ, Rai B, Dorr W, Kirisits C, Bentzen SM, Potter R, Tanderup K; EMBRACE Collaborative Group. Dose-effect relationship and risk factors for vaginal stenosis after definitive radio(chemo)therapy with image-guided brachytherapy for locally advanced cervical cancer in the EMBRACE study. Radiother Oncol. 2016 Jan;118(1):160-6. doi: 10.1016/j.radonc.2015.12.025. Epub 2016 Jan 9. PMID 26780997
- [Background] Sekse RJ, Hufthammer KO, Vika ME. Sexual activity and functioning in women treated for gynaecological cancers. J Clin Nurs. 2017 Feb;26(3-4):400-410. doi: 10.1111/jocn.13407. Epub 2016 Jun 23. PMID 27239803